CLINICAL TRIAL: NCT02738346
Title: Randomized Study Comparing Two Strategies Carboplatin and Etoposide Topotecan in Patients With SCLC on the Second Row With Relapsed at Least Three Months After Initial Response to Chemotherapy With Platinum-etoposide 6 Cycles
Brief Title: SCLC on the 2nd Line With Relapsed After Response to Chemotherapy GFPC 01-2013
Acronym: CBPC
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Angers (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CHU-P 2012-08; GFPC 01-2013 (Other: GFPC)
Record Dates: First submitted 2016-04-04; First posted 2016-04-14 (Estimated); Last update posted 2016-04-25 (Estimated); Status verified 2016-04

CONDITIONS: Small Cell Lung Cancer
Keywords: Small Cell Lung Cancer; Topotecan; Etoposide
MeSH Terms: conditions — Small Cell Lung Carcinoma | interventions — Carboplatin; Etoposide; Topotecan; Tomography, X-Ray Computed

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm A : Carboplatin-Etoposide (Experimental): Intravenous administration of Carboplatin Auc 5 at Day 1 and Intravenous administration of 100 mg / m² / of Etoposide J Day 1 to Day 3 The CT scans evaluations will be conducted during chemotherapy every 6 weeks
  Interventions: Drug: Carboplatin; Drug: Etoposide; Device: CT scans
- Arm B : Topotecan (Active Comparator): Per os administration of 2.3 mg / m² of Topotecan Day 1 to Day 5 The CT scans evaluations will be conducted during chemotherapy every 6 weeks
  Interventions: Drug: Topotecan; Device: CT scans

INTERVENTIONS:
Drug: Carboplatin — Intravenous administration of Carboplatin AUC 5 at Day 1, Every 3 weeks, maximum 6 cycles
  Arms: Arm A : Carboplatin-Etoposide
Drug: Etoposide — Intravenous administration of 100mg/m²/day of Etoposide, Day 1 to Day 3 Every 3 weeks, maximum 6 cycles
  Arms: Arm A : Carboplatin-Etoposide
Drug: Topotecan — Per os administration of 2.3 mg / m2 of Topotecan, Day 1 to Day 5 Every 3 weeks, maximum 6 cycles
  Arms: Arm B : Topotecan
Device: CT scans — The CT scan evaluations will be conducted during chemotherapy every 6 weeks

SUMMARY:
The purpose of this study was to determine prospectively in all patients with SCLC in second line therapy that progression-free survival with the expected reintroduction of platinum / etoposide is greater progression-free survival in the standard arm (topotecan ) in patients who have relapsed at least three months after initial chemotherapy with platinum-etoposide

DETAILED DESCRIPTION:
Topotecan is currently the only drug approved in Europe and the United States for the treatment of second line of SCLC when the recovery first line of treatment is considered inappropriate. This raises the problem of knowing when the recovery first line of treatment should be considered appropriate. Secondly, the effectiveness of response to chemotherapy can be predicted based on the response to initial chemotherapy and the time interval after stopping first line treatment. A complete response after initial treatment and a long disease-free interval are predictors of better response to a second-line treatment. There are two groups: the said patients 'sensitive', which correspond to the first-line chemotherapy and who have relapsed at least 90 days after the first-line treatment and a group of so-called patients "Refractory" refers patients who progress in 90 days or patients who have not responded or progressed during first-line treatment. Median survival is very different depending on whether patients with so-called "sensitive" or "refractory".

When relapse occurs six months after the end of the first line chemotherapy, the usual practice is to reintroduce the first-line treatment. This is based on old studies where the number of patients included was low. If the interval of time after the first line of treatment is ≥ three months, two second-line treatment strategies are possible resumption of initial chemotherapy or topotecan. The combination of cisplatin with etoposide have shown high response rate, whatever the time of relapse. There are, however, no randomized study in the literature comparing topotecan to the reintroduction of a platinum salt associated etoposide.

This study is Randomized, multicenter, controlled, open-label, second line, 2 arms.

Arm A : Carboplatin Auc 5 J1 Etoposide 100 mg / m² / J J1 to J3 IV Arm B : topotecan 2.3 mg / m²J1 to J5 po

1 line by Etoposide Cisplatin or carboplatin etoposide Time interval between the first-line chemotherapy and relapse ≥ 90 days (the date is set at J1 of the last cycle) J-28: TDM thoracoabdominal, brain CT or MRI brain, J 7: Biology, quality of life questionnaire (Lung Cancer Symptom Scale). Assessment of tumor response every 6 weeks during chemotherapy post-chemotherapy followed 2nd line: TDM every 8 weeks until progression or death.

The duration of the participation of each patient included in the trial will be from inclusion through 12 months.

The planned total duration of the trial will be 5 years including 4 years of patient inclusion

ELIGIBILITY:
Inclusion Criteria:

* Lung Cancer Small cell histologically confirmed.
* SCLC stage IV according to the TNM classification in 2009
* Relapse localized SCLC treated with chemoradiotherapy if they are outside the radiation field.
* Patients who have had an objective response to first-line chemotherapy with cisplatin and etoposide or carboplatin and etoposide and have a time interval > or = 90 days between relapse and first-line chemotherapy (the date is set J1 of the last cycle)
* At least one-dimensionally measurable disease (RECIST)
* Age > or = 18 years
* Weight loss <10% during the last 3 months
* Performance status (PS) < or = 2
* Creatinine clearance> 45 ml / min.
* Neutrophils >1,5X10 9 / L and platelets > 100X109 / L.
* Bilirubin < 1,5 X normal.
* Transaminases, alkaline phosphatase < 2,5 X normal except in cases of hepatic metastases (5 X normal).
* Informed Consent signed
* Patients with asymptomatic brain metastases may be included
* Prophylactic brain irradiation based on the habits of each center defined in advance

Exclusion Criteria:

* Lung cancer non-small cell or mixed form (small cell / non-small cell) or absence of histological evidence
* SCLC stage I or stage II or stage III.
* Patients who have not had an objective response to first-line chemotherapy with cisplatin and etoposide or carboplatin and etoposide or that have a time interval < 90 days between relapse and first-line chemotherapy (the date is defined in J1 of the last cycle)
* Serum Na < 125 mmol / L
* Hypercalcemia despite corrective treatment
* Brain metastases or symptomatic meningeal
* A history of malignancy within the last 5 years with the exception of basal cell carcinoma of the skin or carcinoma in situ of the cervix.
* Other concomitant serious medical conditions: congestive heart failure, unstable angina, significant arrhythmia or previous myocardial in the previous six months trial
* Severe or uncontrolled systemic diseases, the investigator found incompatible with the proposed protocol
* Neurological and psychiatric disorders prohibiting comprehension test
* Severe infectious disease during or fever > 38 ° C
* Peripheral neuropathy > or = grade 2
* Any geographical or psychological condition does not allow a proper understanding and compliance with the protocol.
* Private Patient freedom following a judicial or administrative decision
* Pregnant woman, parturient or nursing; Women of childbearing potential and men with a woman of childbearing age must have adequate contraception for the duration of the study and up to 6 months after treatment ends.
* Patient in an exclusion period for another Biomedical study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 164 (Estimated)
Dates: Start 2013-07; Primary Completion 2017-07 (Estimated); Study Completion 2017-07 (Estimated)

PRIMARY OUTCOMES:
Benefit in terms of progression-free survival of a therapeutic strategy | 18 weeks
  Determine the benefit in terms of progression-free survival of a therapeutic strategy by second-line carboplatin etoposide versus topotecan in patients who relapsed at least three months after the initial chemotherapy with platinum-etoposide.

SECONDARY OUTCOMES:
Objective response rate assessed by RECIST | 18 weeks
Overall survival | 18 weeks
Name and number of with treatment-related adverse events as assessed by CTCAE v4.0". | 18 weeks
The quality of life | 18 weeks
  the method of assessment : questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Nathalie BAIZE, Principal Investigator — Angers University Hospital Center
Locations (1):
- Angers University Hospital, Angers, France

REFERENCES:
- [Derived] Baize N, Monnet I, Greillier L, Geier M, Lena H, Janicot H, Vergnenegre A, Crequit J, Lamy R, Auliac JB, Letreut J, Le Caer H, Gervais R, Dansin E, Madroszyk A, Renault PA, Le Garff G, Falchero L, Berard H, Schott R, Saulnier P, Chouaid C; Groupe Francais de Pneumo-Cancerologie 01-13 investigators. Carboplatin plus etoposide versus topotecan as second-line treatment for patients with sensitive relapsed small-cell lung cancer: an open-label, multicentre, randomised, phase 3 trial. Lancet Oncol. 2020 Sep;21(9):1224-1233. doi: 10.1016/S1470-2045(20)30461-7. PMID 32888454